CLINICAL TRIAL: NCT03310983
Title: Growth and Adiposity in Newborns: The Influence of Prenatal Docosahexaenoic Acid (DHA) Supplementation
Acronym: ADORE-GAINS
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00140895
Record Dates: First submitted 2017-10-10; First posted 2017-10-16 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-05

CONDITIONS: Pregnancy; Nutritional Diseases
Keywords: Fat mass; Gestational weight gain; Fetal adipose tissue
MeSH Terms: conditions — Gestational Weight Gain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ADORE- 200 mg/day: Participants enrolled in the ADORE study that were randomly assigned to the 200 mg/day group that consented to participate in ADORE-GAINS.
- ADORE - 1000 mg/day: Participants enrolled in the ADORE study that were randomly assigned to the 1000 mg/day group that consented to participate in ADORE-GAINS.

SUMMARY:
The purpose of this study is to learn if participants in the ADORE study (NCT02626299), who took a DHA supplement during pregnancy, see favorable body fat in their infants from birth to 24 months, and if excessive or appropriate weight gain during pregnancy impacts this result.

ELIGIBILITY:
Participants for this study are invited from the parent study, ADORE. Eligibility listed reflects criteria for the ADORE study.

Inclusion Criteria:

* Agree to consume study capsules and a typical prenatal supplement of 200 mg DHA
* Available by telephone

Exclusion Criteria:

* Expecting multiple infants
* Gestational age at baseline <12 weeks or >20 weeks
* Unable or unwilling to agree to consume capsules until delivery
* Unwilling to discontinue use of another prenatal supplement with DHA that contains ≥ 200 mg DHA
* Women with allergy to any component of DHA product (including algae), soybean oil or corn oil

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are invited from those already participating in the parent study, ADORE.
Sampling Method: Non-Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly Hull, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- The University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Hull HR, Brown A, Gajewski B, Sullivan DK, Carlson SE. The Effect of Prenatal Docosahexaenoic Acid Supplementation on Offspring Fat Mass and Distribution at 24 Months Old. Curr Dev Nutr. 2024 May 11;8(6):103771. doi: 10.1016/j.cdnut.2024.103771. eCollection 2024 Jun. PMID 38948108
- [Derived] Hull HR, Gajewski BJ, Sullivan DK, Carson SE. Growth and adiposity in newborns study (GAINS): The influence of prenatal DHA supplementation protocol. Contemp Clin Trials. 2023 Sep;132:107279. doi: 10.1016/j.cct.2023.107279. Epub 2023 Jul 3. PMID 37406769
- See also: ADORE Clinicaltrials.gov Record - Parent Study — https://clinicaltrials.gov/ct2/show/NCT02626299

RESULTS

PARTICIPANT FLOW:
Groups:
- 200 MG/DAY; 1000 MG/DAY: Docosahexaenoic acid: The main study, ADORE, includes providing DHA to participants during pregnancy. No intervention is included as part of this study.
Period: Overall Study
Arm/Group | 200 MG/DAY | 1000 MG/DAY
Started | 126 | 128
Completed | 111 | 111
Not Completed | 15 | 17
Not completed — Lost to Follow-up | 15 | 17

BASELINE CHARACTERISTICS:
Groups:
- ADORE- 200 mg/Day: Participants enrolled in the ADORE study that were randomly assigned to the 200 mg/day group that consented to participate in ADORE-GAINS.
  200 mg/day Docosahexaenoic acid: The main study, ADORE, includes providing DHA to participants during pregnancy.
- ADORE - 1000 mg/Day: Participants enrolled in the ADORE study that were randomly assigned to the 1000 mg/day group that consented to participate in ADORE-GAINS.
  1000 mg/day Docosahexaenoic acid: The main study, ADORE, includes providing DHA to participants during pregnancy.
- Total: Total of all reporting groups
Arm/Group | ADORE- 200 mg/Day | ADORE - 1000 mg/Day | Total
Number analyzed (Participants) | 126 | 128 | 254
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (5.1) | 31.3 (5.6) | 30.9 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 128 | 254
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Maternal Race and Ethnicity: American Indian or Alaska Native | 1 | 0 | 1
  Maternal Race and Ethnicity: Asian | 0 | 5 | 5
  Maternal Race and Ethnicity: Black or African American | 13 | 10 | 23
  Maternal Race and Ethnicity: Hispanic | 43 | 53 | 96
  Maternal Race and Ethnicity: White | 66 | 59 | 125
  Maternal Race and Ethnicity: More than one race | 3 | 1 | 4
DHA mean % of RBC Total Fatty Acids [Mean (Standard Deviation); unit: percent of total fatty acids in RBC] | 6.5 (1.7) | 6.1 (1.6) | 6.3 (1.6)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.2 (6.9) | 29.1 (8.1) | 28.7 (7.5)

OUTCOME MEASURES:

1. Primary Outcome: Infant Fat Mass (FM)
Description: Difference in FM in offspring exposed to high vs. low DHA and excessive vs. non-excessive GWG
Time Frame: 24 months
Population: Of the participants that completed the 24 month visit, many refused or were uncooperative during the DXA scan. And even a higher percentage were deemed unusable scans due to infant movement.
Measure: Mean (95% Confidence Interval); unit: g
Arm/Group | 200 MG/DAY | 1000 MG/DAY
Number analyzed (Participants) | 31 | 28
g | 3050.7 [2697.3 to 3404.1] | 3673.6 [3248.6 to 4098.7]

2. Secondary Outcome: Central Fat Mass
Description: Difference in FM in offspring exposed to high vs. low DHA and excessive vs. non-excessive GWG
Time Frame: 24 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: g
Arm/Group | 200 MG/DAY | 1000 MG/DAY
Number analyzed (Participants) | 31 | 28
g | 1085.3 [934.3 to 1236.2] | 1377.3 [1195.8 to 1558.8]

ADVERSE EVENTS:
Time Frame: Collected for the duration of study visits, 24 months.
Arm/Group | 200 MG/DAY | 1000 MG/DAY
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/126
Serious Adverse Events (participants affected / at risk) | 0/124 | 0/126
Other Adverse Events (participants affected / at risk) | 0/124 | 0/126

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/83/NCT03310983/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/83/NCT03310983/ICF_001.pdf